CLINICAL TRIAL: NCT06996145
Title: Study of the Isometry of the Anterior Cruciate Ligament From the Center of the Native MRI Insertion Reported on Dynamic Scanner
Acronym: PLANISOLCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2024_843_0104
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament (ACL); Reconstruction; Software
Keywords: anterior cruciate ligament; reconstruction; software; planning; tunnel; isometry; navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dynamic 4D scanner — dynamic 4D scanner

SUMMARY:
In anterior cruciate ligament (ACL) reconstruction, navigation and robotic assistance now provide the possibility of precise positioning of the tunnels.

The challenge is therefore to carry out isometric preoperative planning which can be carried out with robotic or navigation assistance.

In the classic reconstruction technique this isometry is assumed by positioning the tunnels on the center of the native ACL footprints. However, studies cast doubt on this hypothesis.

In this work, the investigators will study the isometry of the center of the native footprints on a dynamic 4D scanner in order to obtain the variation in the distance between the centers of the native footprints during a knee flexion cycle.

This study is part of a larger project. the objective is, if the absence of isometry of the center of the native impressions is confirmed, to develop software assistance which will help the surgeon plan preoperatively an isometric reconstruction. The hypothesis is that the techniques based on the center of the native footprints does not allow isometric reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 or older
* Signed informed consent
* Affiliation to a social security system
* Negative pregnancy test for women of childbearing age

Exclusion Criteria:

* Volunteer having already undergone knee ligament reconstruction or having peri- or intra-articular knee fractures
* Volunteers for whom ligamentoplasty would not have been the therapeutic option chosen in the event of an ACL rupture
* Pregnant woman
* Volunteer under guardianship or curators, under the protection of justice or deprived of public law.
* Minor volunteer
* Contraindication to MRI or scanner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
variation in length of the ACL | 15 days
  Study of the variation in length of the ACL (isometry) during knee flexion in 4D imaging calculated from the center of the natural footprints of the ACL.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No